CLINICAL TRIAL: NCT06568705
Title: Hypofractionated Online Adaptive Radiotherapy of Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HF_BCoART
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Online Adaptive Radiotherapy; Breast Cancer; Hypofractionated Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 26Gy/5f online adaptive radiotherapy (Experimental): The CTV receives a dose of 26Gy in 5 fractions by online adaptive radiotherapy.
  Interventions: Radiation: Ultrafractionated Radiation Treatment
- 43.5Gy/15f online adaptive radiotherapy (Active Comparator): The CTV receives a dose of 43.5Gy in 15 fractions by online adaptive radiotherapy.
  Interventions: Radiation: Moderate hypofractionated Radiation Treatment

INTERVENTIONS:
Radiation: Moderate hypofractionated Radiation Treatment — The online adaptive radiotherapy workflow is used to deliver radiation dose. The CTV of ipsilateral breast receives a dose of 43.5Gy in 15 fractions in patients who underwent breast conserving surgery or mastectomy.
  Arms: 43.5Gy/15f online adaptive radiotherapy
Radiation: Ultrafractionated Radiation Treatment — The online adaptive radiotherapy workflow is used to deliver radiation dose. The CTV of ipsilateral breast receives a dose of 26Gy in 5 fractions in patients who underwent breast conserving surgery or mastectomy.
  Arms: 26Gy/5f online adaptive radiotherapy

SUMMARY:
The goal of this clinical trial is to explore the application of online adaptive radiotherapy in patients who receive moderate hypofractionated or ultrafractionated radiotherapy after breast cancer surgery. The main questions it aims to answer are:

* Can online adaptive radiotherapy improve the accuracy of dose delivery?
* In patients undergoing online adaptive radiotherapy, how are the treatment-related toxicities and tumor control outcomes?

Participants will Receive moderate hypofractionated radiotherapy using online adaptive radiotherapy, a dose of 43.5Gy in 15 fractions or receive ultrafractionated radiotherapy using online adaptive radiotherapy, a dose of 26Gy in 5 fractions.

DETAILED DESCRIPTION:
Online Adaptive Radiotherapy (ART) is an evolution of image-guided radiotherapy that compresses the entire process of image acquisition, plan design, verification, and radiation delivery into approximately 10-30 minutes during which patients do not need to leave the treatment bed. Online ART features rapid image acquisition, automatic contouring and plan optimization supported by artificial intelligence. Body position deviation, breast soft tissue deformation, and organ movement in different treatment fractions can affect the accuracy of radiotherapy for breast cancer patients. Online adaptive radiotherapy is expected to have dosimetric advantages in terms of target coverage and organ-at-risk (OAR) dose reduction, thereby reducing treatment-related side effects while ensuring local tumor control.

Moderate hypofractionation (40-43.5Gy/15-16f/3w) has been shown to achieve equivalent local tumor control and patient survival compared to traditional fractionationated regimens (50Gy/25f/5w), and may even reduce acute and late toxicities. Currently, moderate hypofractionationated radiotherapy has been a first-line recommendation for whole breast irradiation following breast cancer surgery. In addition, the FAST-Forward trial evaluated a shorter regimen, the ultrafractionated whole breast radiotherapy (26Gy/5f/1w) and found that local tumor control and normal tissue toxicity were comparable to the moderate hypofractionationated regimen. The Royal College of Radiologists (RCR) has endorsed 5-fraction ultrafractionationated radiotherapy as a standard option for postoperative breast cancer radiation treatment in 2020.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥35 years, <70 years
* ECOG score: 0-2
* Having underwent breast-conserving surgery or Modified radical mastectomy with or without sentinel lymph node biopsy or axillary lymph node dissection
* Pathologically confirmed primary breast cancer
* For patients who did not receive neoadjuvant therapy: pathological staged pT0-2N0-1; for patients who received neoadjuvant therapy: staged ypT0-2N0-1
* Indicated for postoperative adjuvant radiotherapy, planned to undergo postoperative adjuvant radiotherapy
* Able to cooperate and tolerate the treatment

Exclusion Criteria:

* Pathologically confirmed metastasis in supraclavicular or infraclavicular lymph nodes, or distant metastasis
* History of radiotherapy to the neck or chest
* Contraindications or intolerance to radiation therapy (such as pregnancy or lactation, severe impairment of heart, lung, kidney, liver, or other vital organ functions; severe infection or hematologic abnormalities; brachial plexus nerve injury on the affected side; active connective tissue diseases, etc.)
* History of malignant tumors

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The dose coverage of target volume as assessed by planning tumor volume V100% | 3 months after radiotherapy
  Planning tumor volume V100%, defined as the planning tumor volume receiving at least 100% of the prescribed dose (V100%), is used to evaluate the dose coverage of target volume.

SECONDARY OUTCOMES:
Treatment-related toxicity | Baseline; Every week during radiotherapy; 1 week, 2 weeks, 3/6/12/24 months after radiotherapy.
  Toxicity is evaluated by Common Terminology Criteria for Adverse Events v5.0.
Local recurrence rate (LRR) | 3, 6, 12, 24 months after radiotherapy
  LRR will be deducted from the local recurrence survival defined as the interval between date of surgery and the occurrence of local relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China